CLINICAL TRIAL: NCT04649749
Title: Central Programming in Patients With a Bionic Hand After Traumatic Brachial Plexus Injury
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Galia Valentinova Anguelova, Visiting Researcher at Medical University of Vienna, Austria, Medical University of Vienna
Other Study IDs: 1955/2020
Record Dates: First submitted 2020-10-01; First posted 2020-12-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Brachial Plexus Neuropathies; Traumatic Brachial Plexus Lesion; Bionic Hand Reconstruction
Keywords: traumatic brachial plexus lesion; bionic hand reconstruction; hand amputation; hand prosthesis; central programming; fMRI; resting state networks; DTI
MeSH Terms: conditions — Brachial Plexus Neuropathies | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients - bionic hand acquired: 3 adult patients who acquired a bionic hand at the Medical University of Vienna after a traumatic brachial plexus lesion.
  Interventions: Diagnostic Test: MRI
- Patients - bionic hand not yet acquired: 3 patients eligible for the bionic hand prior to a possible amputation.
  Interventions: Diagnostic Test: MRI
- Control subjects: Ten control subjects will be included for comparison.
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI scan
  Other Names: functional MRI; fMRI

SUMMARY:
Traumatic brachial plexus lesions may lead to permanent impairment of hand function despite brachial plexus surgery. In selected cases the affected forearm can be amputated and replaced by a bionic hand. It is unclear how cortical activation patterns change after the injury and after acquisition of the hand prosthesis considering the complex changes in sensory and motor feedback. The aim of the study is to measure cortical activity with fMRI during actual and imagery movements with the affected and healthy arm in a group of patients after traumatic brachial plexus injury and a group in whom this was followed by replacement with a bionic hand. In this prospective study three groups of patients will participate: 1) 3 adult patients with a traumatic brachial plexus lesion eligible for a bionic arm but prior to its acquisition, 2) 3 patients with a traumatic brachial plexus lesion who have acquired the bionic arm already, and 3) 10 healthy subjects. The investigators will measure cortical activity using fMRI BOLD tasks of closing the hand and motor imagery of this movement. Cortical activity will be compared between the three groups. Additionally, regional gray matter volume, resting-state, and DTI networks will be studied. Written informed consent will be provided prior to the investigation. The complete examination has a duration of approximately 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* participants should understand German or English
* patients with a bionic hand are selected who are able to open and close the hand prosthesis.

Exclusion Criteria:

* the standard contraindications for MRI will be checked for according to hospital protocol (ferromagnetic devices such as clips, claustrophobia, etc.) and, if necessary, patients will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of 3 adult patients who acquired a bionic hand at the Medical University of Vienna after a traumatic brachial plexus lesion, and a group of 3 patients eligible for the bionic hand prior to a possible amputation will be included. The number of patients included is based on the rarity of the procedure and thus the very limited number of eligible study participants. Ten control subjects will be included for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
task-related cortical activity - fMRI BOLD signal | MRI task scanning approximately 20 minutes
  The investigators will measure cortical activity measured as a fMRI BOLD (blood-oxygen-level-dependent) signal, during four tasks: closing the hand (lef tand right) and motor imagery of this movement.

SECONDARY OUTCOMES:
resting state activity - fMRI BOLD signal | MRI resting state scanning approximately 10 minutes
  The investigators will measure brain activity measured as a fMRI BOLD signal (blood-oxygen-level-dependent) during rest.
diffusion tensor imaging (DTI) MRI | DTI scanning approximately 10 minutes
  The investigators will measure mean diffusivity of the brain with DTI.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Aszmann, prof. dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aszmann OC, Roche AD, Salminger S, Paternostro-Sluga T, Herceg M, Sturma A, Hofer C, Farina D. Bionic reconstruction to restore hand function after brachial plexus injury: a case series of three patients. Lancet. 2015 May 30;385(9983):2183-9. doi: 10.1016/S0140-6736(14)61776-1. Epub 2015 Feb 25. PMID 25724529
- [Background] Sturma A, Hruby LA, Prahm C, Mayer JA, Aszmann OC. Rehabilitation of Upper Extremity Nerve Injuries Using Surface EMG Biofeedback: Protocols for Clinical Application. Front Neurosci. 2018 Dec 4;12:906. doi: 10.3389/fnins.2018.00906. eCollection 2018. PMID 30564090
- [Background] Decety J, Grezes J. Neural mechanisms subserving the perception of human actions. Trends Cogn Sci. 1999 May;3(5):172-178. doi: 10.1016/s1364-6613(99)01312-1. PMID 10322473
- [Background] Lotze M, Flor H, Grodd W, Larbig W, Birbaumer N. Phantom movements and pain. An fMRI study in upper limb amputees. Brain. 2001 Nov;124(Pt 11):2268-77. doi: 10.1093/brain/124.11.2268. PMID 11673327
- [Background] Hotz-Boendermaker S, Funk M, Summers P, Brugger P, Hepp-Reymond MC, Curt A, Kollias SS. Preservation of motor programs in paraplegics as demonstrated by attempted and imagined foot movements. Neuroimage. 2008 Jan 1;39(1):383-94. doi: 10.1016/j.neuroimage.2007.07.065. Epub 2007 Aug 23. PMID 17919932
- [Background] Date S, Kurumadani H, Yoshimura M, Fukae A, Onishi K, Hayashi J, Shinomiya R, Sunagawa T. Long-term disuse of the hand affects motor imagery ability in patients with complete brachial plexus palsy. Neuroreport. 2019 Apr 10;30(6):452-456. doi: 10.1097/WNR.0000000000001229. PMID 30855560
- [Background] Anguelova GV, Rombouts SARB, van Dijk JG, Buur PF, Malessy MJA. Increased brain activation during motor imagery suggests central abnormality in Neonatal Brachial Plexus Palsy. Neurosci Res. 2017 Oct;123:19-26. doi: 10.1016/j.neures.2017.05.001. Epub 2017 May 4. PMID 28479130

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04649749/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT04649749/ICF_000.pdf